CLINICAL TRIAL: NCT07007949
Title: Ivosidenib Combined With Venetoclax and Azacitidine for the Treatment of Newly Diagnosed IDH1 Mutation Acute Myeloid Leukemia: a Prospective, Single-arm, Two-cohorts, Study
Brief Title: a New Treatment of Newly Diagnosed IDH1 Mutation Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Prof., The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVO01
Record Dates: First submitted 2025-05-09; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; IDH1 Gene Mutation; Ivosidenib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unfit Arm (Experimental): Unfit subjects should be treated for a minimum of 6 cycles of combination therapy unless they experience relapse after achieving a CR, CRi (including CRp), or morphologic leukemia-free state (MLFS); disease progression after having previously attained partial remission (PR) or stable disease; unacceptable toxicity (adverse event [AE]); confirmed pregnancy; withdrawal by subject; protocol violation; death; end of Study or other Protocol-specified event endpoints (refer to study design).
  Interventions: Drug: Ivosidenib combined with venetoclax and azacitidine
- Fit Arm (Experimental): Fit subjects should be treated for a minimum of 2 cycles of combination therapy unless they experience relapse after achieving a CR, CRi (including CRp), or morphologic leukemia-free state (MLFS); disease progression after having previously attained partial remission (PR) or stable disease; unacceptable toxicity (adverse event [AE]); confirmed pregnancy; withdrawal by subject; protocol violation; death; end of Study or other Protocol-specified event endpoints (refer to study design).
  Interventions: Drug: Ivosidenib combined with venetoclax and azacitidine

INTERVENTIONS:
Drug: Ivosidenib combined with venetoclax and azacitidine — • Ivosidenib (Ivo): The dosage is 500 mg, administered orally once daily (QD). Oral administration begins on Day 15 of Cycle 1 (C1D15) and continues on each subsequent day of the following cycles. Each cycle lasts 28 days (±2 days), with continuous dosing. • Venetoclax (Ven): The dosage is 100 mg on Day 1 of Cycle 1 (C1D1), 200 mg on Day 2 of Cycle 1 (C1D2), and 400 mg on Days 3-14 of Cycle 1 (C1D3-14), administered orally once daily (QD). For subsequent cycles, the dosage is 400 mg on Days 1-14, administered orally once daily (QD). • Azacitidine (Aza): The dosage is 75 mg/m² per day, administered via subcutaneous injection (Subcutaneous injection, SC) or intravenous injection (Intravenous, IV). It is given during the first week (7 days) of each 4-week (28-day) cycle (or according to the 5-2-2 dosing schedule). Whenever possible, each subject should use the same dosing schedule throughout the treatment period.
  Other Names: Unfit Arm
  Arms: Unfit Arm
Drug: Ivosidenib combined with venetoclax and azacitidine — • Ivosidenib (Ivo): The dosage is 500 mg, administered orally once daily (QD). Oral administration begins on Day 15 of Cycle 1 (C1D15) and continues on each subsequent day of the following cycles. Each cycle lasts 28 days (±2 days), with continuous dosing. • Venetoclax (Ven): The dosage is 100 mg on Day 1 of Cycle 1 (C1D1), 200 mg on Day 2 of Cycle 1 (C1D2), and 400 mg on Days 3-14 of Cycle 1 (C1D3-14), administered orally once daily (QD). For subsequent cycles, the dosage is 400 mg on Days 1-14, administered orally once daily (QD). • Azacitidine (Aza): The dosage is 75 mg/m² per day, administered via subcutaneous injection (Subcutaneous injection, SC) or intravenous injection (Intravenous, IV). It is given during the first week (7 days) of each 4-week (28-day) cycle (or according to the 5-2-2 dosing schedule). Whenever possible, each subject should use the same dosing schedule throughout the treatment period.
  Other Names: Fit Arm
  Arms: Fit Arm

SUMMARY:
This is a single arm, open-label, multicenter clinical trial to evaluate the efficacy and safety of ivosidenib+venetoclax+ azacitidine in adult Chinese subjects with newly diagnosed IDH1m AML.A total of approximately 42 China Nationwide subjects with newly diagnosed IDH1m AML will participate in the study.The primary endpoint of the study is the complete remission(CR) + CR with partial hematologic recovery(CRh) rate, and the key secondary endpoints are CR rate,event-free survival (EFS),overall survival (OS),the objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age
2. Have previously untreated AML, defined according to World Health Organization criteria. Subjects with extramedullary disease alone (ie, no detectable bone marrow and no detectable peripheral blood AML) are not eligible for the study.
3. Have an IDHl mutation resulting in an R132C, R132G, R132H, R132L, or R132S substitution.
4. Have an ECOG PS score of 0 to 2.
5. Have adequate hepatic function, as evidenced by:

   * Serum total bilirubin ≤2 × ULN, unless considered to be due to Gilbert's disease or underlying leukemia, where it must be <3 x ULN.
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤3.0 × ULN, unless considered to be due to underlying leukemia.
6. Have adequate renal function, as evidenced by serum creatinine ≤2.0 x ULN or creatinine clearance >30 mL/min based on the Cockcroft-Gault glomerular filtration rate.
7. Have agreed to undergo serial blood and bone marrow sampling.
8. Be able to understand and willing to sign an informed consent form.
9. Be willing to complete QoL assessments during study treatment and at the designated time points following treatment discontinuation.
10. If female with reproductive potential, must have a negative serum pregnancy test prior to the start of study therapy. Female subjects with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion or who have not been naturally postmenopausal for at least 24 consecutive months. Females of reproductive potential, as well as fertile men with female partners of reproductive potential, must use 2 effective forms of contraception (including at least 1 barrier form) from the time of giving informed consent throughout the study and for 90 days (both females and males) following the last dose of study drugs). Effective forms of contraception are defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal ligation, condoms with spermicide, or male partner sterilization.

Exclusion Criteria:

1. Have received any prior treatment for AML with the exception of nononcolytic treatments to stabilize disease such as hydroxyurea or leukapheresis.
2. Have received a hypomethylating agent for myelodysplastic syndrome (MDS).
3. Subject has favorable risk cytogenetics such as t(8;21), inv(16), t(16;16) or t(15;17).
4. Subject has acute promyelocytic leukemia
5. Subjects who had previously received treatment for an antecedent hematologic disorder, including investigational agents, may not be randomized until a washout period of at least 5 half-lives of the investigational agent has elapsed since the last dose of that agent.
6. Have received prior treatment with an IDH1 inhibitor or BCL-2 inhibitor.
7. Have a known hypersensitivity to any of the components of Ivosidenib, venetoclax, or azacitidine.
8. Are female and pregnant or breastfeeding.
9. Are taking known strong cytochrome P450 (CYP) 3A4 inducers or sensitive CYP3А4 substrate medications with a narrow therapeutic window, unless they can be transferred to other medications within ≥5 half-lives prior to dosing.
10. Have an active, uncontrolled, systemic fungal, bacterial, or viral infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
11. Have a prior history of malignancy other than MDS or myeloproliferative disorder, unless the subject has been free of the disease for ≥1 year prior to the start of study treatment. However, subjects with the following history/concurrent conditions or similar indolent cancer are allowed to participate in the study:

    * Basal or squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
12. Have had significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association Class (NYHA) Class III or IV congestive heart failure, myocardial infarction, unstable angina, and/or stroke.
13. Have a heart-rate corrected QT interval using Fridericia's method (QTcF) >470 msec or any other factor that increases the risk of QT prolongation or arrhythmic events (eg, NYHA Class III or IV congestive heart failure, hypokalemia, family history of long QT interval syndrome). Subjects with prolonged QTcF interval in the setting of bundle branch block may participate in the study.
14. Have a known infection caused by human immunodeficiency virus or active hepatitis B virus (HBV) or hepatitis C virus that cannot be controlled by treatment.
15. Have dysphagia, short-gut syndrome, gastroparesis, or any other condition that limits the ingestion or gastrointestinal absorption of orally administered drugs.
16. Have uncontrolled hypertension (systolic blood pressure [BP] >180 mmHg or diastolic BP>100 mmHg).
17. Have clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid during Screening is only required if there is a clinical suspicion of CNS involvement by leukemia during Screening.
18. Have immediate, life-threatening, severe complications of leukemia, such as uncontrolled bleeding, pneumonia with hypoxia or sepsis, and/or disseminated intravascular coagulation.
19. Have any other medical or psychological condition deemed by the Investigator to be likely to interfere with the subject's ability to give informed consent or participate in the study.
20. Are taking medications that are known to prolong the QT interval unless they can be transferred to other medications within ≥5 half-lives prior to dosing, or unless the medications can be properly monitored during the study. (If equivalent medication is not available, heart rate corrected QT interval [QTc] will be closely monitored.)
21. Subjects with a known medical history of progressive multifocal leukoencephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CR + CRh rate | 1 year
  CR is defined as Bone marrow blasts <5% and no Auer rods; absence of extramedullary disease; ANC ≥1.0 × 109/L (1000/µL); platelet count ≥100 × 109/L (100,000/µL); independence of red blood cell transfusions.
  CRh is defined as a CR with partial recovery of peripheral blood counts where absolute neutrophil count (ANC) is > 0.5 × 109/L [500/µL], and platelet count is > 50 × 109/L [50,000/µL].

SECONDARY OUTCOMES:
CR rate | 1 year
  CR is defined as bone marrow blasts < 5% and no Auer rods, absence of extramedullary disease, ANC ≥ 1.0 × 109/L [1000/µL], platelet count ≥ 100 × 109/L [100,000/µL], and independence of RBC transfusions).
EFS | 1 year
  Event-free survival (EFS) is defined as the time from Cycle 1, Day 1 (C1D1) until treatment failure, relapse from remission, or death from any cause, whichever occurs first. Treatment failure is defined as failure to achieve CR by Week 24.
OS | 1 year
  Overall survival (OS) is defined as the time from date of C1D1 to the date of death due to any cause.
ORR | 1 year
  Objective response rate (ORR) is defined as the rate of CR, CRi (including complete remission with incomplete platelet recovery [CRp], PR, and MLFS.

OTHER OUTCOMES:
CR + CRi (including CRp) rate | 1 year
  CR is defined as Bone marrow blasts <5% and no Auer rods; absence of extramedullary disease; ANC ≥1.0 × 109/L (1000/µL); platelet count ≥100 × 109/L (100,000/µL); independence of red blood cell transfusions.
  CRi (including CRp) is defined as all CR criteria except for residual neutropenia (ANC <1.0 × 109/L [1000/µL]) or thrombocytopenia (platelet counts <100 × 109/L [100,000/µL]; without platelet transfusion for at least 1 week prior to disease assessment).
DOCR，DOCRh，DOR，DOCRi | 1 year
  DOCR, among subjects who achieved CR; DOCRh, among subjects who achieved CR or CRh; DOR, among subjects who achieved CR, CRi (including CRp), PR, and/or MLFS; and DOCRi, among subjects who achieved CR or CRi (including CRp).
  MLFS is defined as bone marrow blasts <5% and no Auer rods; absence of extramedullary disease; no hematologic recovery required.
  PR is defined as all hematologic criteria of CR; decrease of bone marrow blast percentage to 5%-25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
TTCR，TTCRh，TTR，TTCRi | 1 year
  TTCR, among subjects who achieved CR; TTCRh, among subjects who achieved CR or CRh; TTR, among subjects who achieved CR, CRi (including CRp), PR, and/or MLFS; and TTCRi, among subjects who achieved CR or CRi (including CRp).
  MLFS is defined as bone marrow blasts <5% and no Auer rods; absence of extramedullary disease; no hematologic recovery required.
  PR is defined as all hematologic criteria of CR; decrease of bone marrow blast percentage to 5%-25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
MRD negativity rate. | 1 year
  To evaluate the measurable residual disease (MRD) negativity rate.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China